CLINICAL TRIAL: NCT00407888
Title: Adjuvant Therapy for High-Risk Localized Breast Cancer Using Weekly Adriamycin + Daily Oral Cytoxan With Continuous G-CSF Support for 12 Weeks Followed by Weekly Abraxane™ for 12 Weeks With Concurrent Herceptin for Subjects With HER-2/Neu Positive Disease, Phase II
Brief Title: Doxorubicin Hydrochloride, Cyclophosphamide, and Filgrastim Followed By Paclitaxel Albumin-Stabilized Nanoparticle Formulation With or Without Trastuzumab in Treating Patients With Breast Cancer Previously Treated With Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Vijayakrishna Gadi, Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6141; NCI-2010-02117 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Estrogen Receptor-positive Breast Cancer; HER2-positive Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor; Taxes; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (Experimental): Patients receive dose-intensive chemotherapy comprising doxorubicin hydrochloride IV over 10-15 minutes on day 1, oral cyclophosphamide once daily on days 1-7, and filgrastim subcutaneously on days 2-7. Courses repeat every 7 days for up to 12 weeks in the absence of disease progression or unacceptable toxicity. Beginning 1 week later, patients then receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes once a week for 12 weeks in the absence of disease progression or unacceptable toxicity. Patients with HER-2/neu positive disease also receive trastuzumab IV over 30-90 minutes once a week for 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: doxorubicin hydrochloride; Drug: cyclophosphamide; Biological: filgrastim; Drug: paclitaxel albumin-stabilized nanoparticle formulation; Biological: trastuzumab; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: cyclophosphamide — Given orally
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Drug: paclitaxel albumin-stabilized nanoparticle formulation — Given IV
  Other Names: ABI-007; nab paclitaxel; nab-paclitaxel; nanoparticle albumin-bound paclitaxel
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
Other: laboratory biomarker analysis — Correlative studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin hydrochloride, cyclophosphamide, and paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Colony-stimulating factors, such as filgrastim, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving combination chemotherapy and filgrastim together with trastuzumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving doxorubicin hydrochloride, cyclophosphamide, and filgrastim together followed by paclitaxel albumin-stabilized nanoparticle formulation and trastuzumab works in treating patients with breast cancer previously treated with surgery

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess disease-free survival following a dose-intensive weekly regimen of Adriamycin + oral cyclophosphamide augmented with G-CSF support followed by Abraxane and Herceptin if appropriate for adjuvant treatment of high risk breast cancer patients.

SECONDARY OBJECTIVES:

I. To assess the toxicity associated with this regimen. II. To assess the delivered dose intensity of the regimen. III. To assess time to treatment failure and overall survival of the regimen. IV. To assess the incidence and severity of delayed nausea and vomiting with this regimen.

OUTLINE:

Patients receive dose-intensive chemotherapy comprising doxorubicin hydrochloride IV over 10-15 minutes on day 1, oral cyclophosphamide once daily on days 1-7, and filgrastim subcutaneously on days 2-7. Courses repeat every 7 days for up to 12 weeks in the absence of disease progression or unacceptable toxicity. Beginning 1 week later, patients then receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes once a week for 12 weeks in the absence of disease progression or unacceptable toxicity. Patients with HER-2/neu positive disease also receive trastuzumab IV over 30-90 minutes once a week for 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically confirmed diagnosis of primary breast carcinoma that has been surgically resected; (this regimen is not intended for neoadjuvant treatment)
* 4 + nodes
* OR if 1-3 + nodes, either ER OR HER-2/neu+
* OR have high-risk node negative disease that is HER-2/neu positive OR >= 2.0 cm tumor size
* HER-2/new + definition: patient has known tumor HER-2/new expression = 3+ by IHC or, if 2+ by IHC confirmed to be FISH positive
* Patients with clinically apparent cardiac disease, or history of same, are not eligible; patients who are >= 60 years of age or who have a history of hypertension must have an echocardiogram or MUGA prior to enrollment; patients with breast cancer that is HER-2/neu positive and a treatment plan that includes Herceptin must have an echocardiogram or MUGA scan prior to enrollment; the LVEF must be within the institutional normal range; if LVEF is > 75%, the investigator should consider having the LVEF reviewed or repeating the MUGA prior to registration
* WBC >= 4,000
* ANC >= 1,500
* Platelet count >= 100,000
* Serum creatinine =< 1.5 x IULN
* Bilirubin =< 2.0
* SGOT/SGPT/alkaline phosphatase =< 2 x IULN
* Elevations greater than these require metastatic work up
* Be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study specific screening procedures

Exclusion Criteria:

* Except for the following, no other malignancy is allowed: synchronous ipsilateral breast cancer of the same subtype (ER/PR, HER-2/neu), adequately treated basal cell or squamous cell skin cancer, in situcervical cancer or other stage I or II cancer from which the patient has been disease free for at least 5 years
* Patients with cardiac disease that would preclude the use of Adriamycin, Taxol or Herceptin are not eligible; this includes:
* Angina pectoris that requires the use of antianginal medication
* Cardiac arrhythmia requiring medication
* Severe conduction abnormality
* Clinically significant valvular disease
* Cardiomegaly on chest x-ray
* Ventricular hypertrophy on EKG
* Uncontrolled hypertension, (diastolic greater than 100 mm/Hg or systolic > 200 mm/hg)
* Current use of digitalis or beta blockers for CHF
* Clinically significant pericardial effusion
* Myocardial infarction documented as a clinical diagnosis or by EKG or any other test
* Documented congestive heart failure
* Documented cardiomyopathy
* Documented arrhythmia or cardiac valvular disease that requires medication or is medically significant
* Patients who have received prior chemotherapy or radiotherapy are not eligible
* Patients who are pregnant or breastfeeding are not eligible; women of child bearing potential must agree to practice adequate contraception
* Patients with active infection are not eligible
* Patients who are known to be infected with HIV, hepatitis B or hepatitis C are not eligible; testing is not required unless there is a high index of clinical suspicion
* Patients suffering from psychiatric impairment are not eligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-05; Primary Completion 2009-05 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vijayakrishna K Gadi, MDPHD, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 52 [29 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 51
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival Following a Dose-intensive Weekly Regimen of Adriamycin + Oral Cyclophosphamide Augmented With G-CSF Support Followed by Abraxane and Herceptin
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 60
Participants | 56

2. Secondary Outcome: Delivered Dose Intensity of the Regimen
Time Frame: After at least one course of Adriamycin, up to 12 weeks.
Measure: Number; unit: percentage of mean administered dose
Arm/Group | Arm I
Number analyzed (Participants) | 60
percentage of mean administered dose
  Doxorubicin | 92.6
  Cyclophosphamide | 92.1
  nP (intent-to-treat) | 88.0

3. Secondary Outcome: Toxicity Associated With This Regimen
Time Frame: After at least one course of Adriamycin, up to 12 weeks.
Population: Some results reported are only considered amongst patients receiving Trastuzumab (n = 15).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 60
Participants
  Filgrastim used | 37
  Dose holds/reductions | 43
  Hospitalization/ER evaluation | 5
  Trastuzumab patients with decease in LVEF to <50%: number analyzed (Participants) | 15
  Trastuzumab patients with decease in LVEF to <50% | 2
  Trastuzumab patients with decease in LVEF to <10%: number analyzed (Participants) | 15
  Trastuzumab patients with decease in LVEF to <10% | 3

4. Secondary Outcome: Time to Treatment Failure
Description: Median time from date of start of therapy to date of removal from therapy for reason other than completion, date of first observation of recurrent disease or date of death due to any cause whichever comes first.
Time Frame: Up to 6 years
Population: Outcome measure reported only for those that had an event (death, recurrent disease or removal).
Measure: Median (Full Range); unit: years
Arm/Group | Arm I
Number analyzed (Participants) | 11
years | 2.7 [0.2 to 4.2]

5. Secondary Outcome: Overall Survival
Description: Count of surviving patients at two years and six years
Time Frame: Up to 6 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 60
Participants
  Two years | 59
  Six years | 53

ADVERSE EVENTS:
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 5/60
Other Adverse Events (participants affected / at risk) | 33/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=60)
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Possible Pneumoncystis Pneumonia (Infections and infestations) | 1
Pneumothorax due to MVA (Respiratory, thoracic and mediastinal disorders) | 1
Febrile Neutopenia (Blood and lymphatic system disorders) | 1
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1
Mucositis (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=60)
Neutropenia (Investigations) | 33
Nausea (Gastrointestinal disorders) | 3
Leukopenia (Investigations) | 3
Low Hemoglobin (Renal and urinary disorders) | 3
Neuropathy (Nervous system disorders) | 4
Mucositis (Gastrointestinal disorders) | 6
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes